CLINICAL TRIAL: NCT02496429
Title: ESP Evaluation of the Reliability and Usability of the Reusable "BrownieForSymphony" Pump Set
Brief Title: Evaluation of the Reliability and Usability of the Reusable "BrownieForSymphony" Pump Set
Acronym: ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MBF1502
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BrownieForSymphony use (Other): Each participant will use the BrownieForSymphony pumpset
  Interventions: Device: BrownieForSymphony use

INTERVENTIONS:
Device: BrownieForSymphony use — Professional will use the BrownieForSymphony Pumpset in their daily work. hospitalized lactating woman will pump with the BrownieForSymphony Pumpset

SUMMARY:
The primary objectives of this study is to evaluate how professionals rate the reliability and usability of the reusable BrownieForSymphony pump set.and the current used Symphony pump set

4.2 Secondary Objectives

The secondary objectives of this study are:

* to evaluate the rate of usability problems with the BrownieForSymphony pump set
* to evaluate the pragmatic quality (task/goal fulfilment) of the BrownieForSymphony pump set
* to evaluate first impression of lactating woman regarding pumping with the BrownieForSymphony pump set

DETAILED DESCRIPTION:
This is a 5 day case study to evaluate the reliability and usability of the BrownieForSymphony pump set.

The study consists of two different participant groups, professionals (e.g. lactation consultants, nurses) and lactating women.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized lactating woman >18 years which are pumping breast milk

Exclusion Criteria:

* hospitalized lactating woman has a medical indication for pumping (e.g. Mastitis, cracked nipples) lactating woman used a breast shield size >27 and <24

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Usability Scale (SUS) Symphony Pumpset usability | day at inclusion
  Rating of the Usability of the Symphony Pumpset
Usability Scale (SUS) BrownieForSymphony Pumpset usability | after 5 days
  Rating of the Usability of the BrownieForSymphony Pumpset

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Prime, PhD, Principal Investigator — Medela AG
Locations (2):
- Germany (2):
  - Klinik Dr. Geißenhofer, Munich
  - University Tuebingen, Tübingen